CLINICAL TRIAL: NCT05673759
Title: The Clinical Utility of ERPs in the Diagnosis of Cognitive Impairment
Brief Title: Event-Related Potential (ERP) Components in Clinical Diagnosis
Status: Terminated | Type: Observational
Why Stopped: The sponsor stopped funding the study.
Sponsor: Boston University (Other)
Collaborators: VoxNeuro Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: H-43360
Record Dates: First submitted 2022-12-07; First posted 2023-01-06 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease; Dementia, Mild; Mild Cognitive Impairment
Keywords: Memory Strategies; EEG headgear; Event-Related Potentials
MeSH Terms: conditions — Alzheimer Disease; Dementia; Lymphoma, Follicular; Cognitive Dysfunction | interventions — Electroencephalography; Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- 75 Mild AD: 75 patients diagnosed with Mild Alzheimer's disease.
  Interventions: Device: Electroencephalogram (EEG) system; Behavioral: Standard Neuropsychological Testing
- 75 MCI due to any etiology: 75 patients diagnosed with Mild Cognitive Impairment due to any etiology.
  Interventions: Device: Electroencephalogram (EEG) system; Behavioral: Standard Neuropsychological Testing
- 25 Healthy Older Adults: 25 Healthy older adults age: 50-90 (control).
  Interventions: Device: Electroencephalogram (EEG) system; Behavioral: Standard Neuropsychological Testing
- 25 Healthy Younger Adults: 25 Healthy younger adults age: 20-50 (control).
  Interventions: Device: Electroencephalogram (EEG) system; Behavioral: Standard Neuropsychological Testing; Behavioral: Additional neuropsychological tests

INTERVENTIONS:
Device: Electroencephalogram (EEG) system — An FDA 510(k) approved EEG/ERP device designed by G-Tec ™ intended for the acquisition, display, analysis, storage, reporting and management of EEG and auditory evoked potentials (AEP) information and uses Bluetooth technology to securely transmit EEG signals to a computer. The device is patient-friendly, and no serious adverse events have occurred to-date in any research or clinical study or in clinical use.
  Other Names: g.Nautilus PRO (G-Tec ™)
Behavioral: Standard Neuropsychological Testing — Prior to the EEG session, neuropsychological testing will be done to establish a baseline measurement. We administer a full standard neuropsychological battery (45 mins) for all participants which includes the following tests: MOCA (only for older participants), MMSE, CERAD, Phonemic Test and the Category Fluency test, Trails Making Test A and B, BNT, BAI, BDI, PANAS, Ishihara Color Blindness test, and the Snellen Eye Chart.
  Other Names: Neuropsychological Battery
Behavioral: Additional neuropsychological tests — Younger participants will receive additional testing along with the standard neuropsychological battery including Pittsburgh Sleep Quality Index (PSQI) [37] for sleep quality measures, the Test of Memory Malingering (TOMM) for effort measure, Ohio State Traumatic Brain Injury Identification Method questionnaire (OSU-TBI) [38] to gather lifetime TBI history, and the Neurobehavioral Symptom Inventory (NBSI) [39] for post-concussive symptoms. These additional tests will add an extra fifteen minutes, making the total time for neuropsychological questionnaires 1 hour in younger participants.
  Groups: 25 Healthy Younger Adults

SUMMARY:
In this study, the investigators will use a novel electroencephalogram (EEG) system that participants will wear during a single in-person research session to investigate whether ERPs are now ready for validation as a tool clinicians can easily implement to increase diagnostic accuracy and confidence. This EEG will not be used to treat, cure, mitigate or diagnosis any disease and there will be no safety or efficacy data collected about the machine for any purpose including support of FDA submission.

The investigators will compare the ERP data to that of neuropsychological testing in order to determine the degree of correlation between these two measures. Questionnaires on cognition, mood, and fluency will be administered prior to the EEG to establish a baseline. ERP data from the EEG session will be compared with the results of the neuropsychological battery in order to determine whether the implementation of ERPs in the existing workflow of clinicians can aid in diagnostic accuracy, thus altering clinical management.

DETAILED DESCRIPTION:
A cross sectional cohort study design with four groups will be implemented to determine how ERPs can provide diagnostic information and alter clinical management beyond that of neuropsychological testing alone in patients with Alzheimer's disease (AD) or Mild Cognitive Impairment (MCI).

Secondary Objectives:

* To determine the impact of ERP testing (using cognitive health assessment reports) on change in research grade clinical diagnosis
* To determine the degree of correlation between quantitative ERP measures with neuropsychological testing performance using a standardized neuropsychological battery.

  75 mild AD dementia and 75 MCI due to any etiology, 25 Older Adults (OA) and 25 Younger Adults (YA) will be enrolled over the course of two years. Each subject will participate in the study for 1 visit.

The in person 50-60-minute testing session consists of a neuropsychological battery, and an EEG session with computer tasks including the Auditory Oddball paradigm, a Continuous Visual Memory Test, Auditory Evoked Potentials, Visual Evoked Potentials, the Erikson Flanker Task, and the Hayling Task.

ELIGIBILITY:
Inclusion Criteria:

For Mild Alzheimer Disease (AD) dementia

* Meets probable AD dementia National Institute on Aging and Alzheimer's Association (NIA-AA) criteria
* 50-90 years old
* Mini-Mental State Examination (MMSE) 20-27
* Performance on delayed recall and recognition memory worse than 1.5 standard deviation (SD) for age and education
* Performance on delayed recall and recognition memory worse than 1.5 SD for age & education in at least one other cognitive domain (e.g., language, executive functioning) based on other tests in our neuropsychological test battery.
* Dr. Turk and Dr. Budson will confirm all mild AD dementia diagnoses

For Mild cognitive impairment (MCI)

* MCI due to any etiology 50-90 years old
* MMSE > 23
* Performance on delayed recall and recognition memory worse than 1.0 SD for age & education adjusted norms
* Dr. Turk and Dr. Budson will confirm all MCI diagnoses

For Healthy older adults

* 50-90 years old
* Functioning normally in occupation determined by self-report

For Healthy younger adults

* 20-50 years old
* Functioning normally in occupation determined by self-report

Exclusion Criteria:

A clinically significant problem of any of the following conditions:

* depression
* heavy alcohol or drug use
* cerebrovascular disease
* a different degenerative disease (e.g., fronto-temporal dementia, Parkinson's disease)
* any medical condition whose severity could significantly impair cognition (e.g., organ failure)
* on any antipsychotic or epilepsy medication
* Unable to understand the consent form

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any participant age: 20-90 years old, with or without a diagnosis of AD or cognitive impairment.
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Electroencephalogram (EEG) memory diagnosis | baseline
  The EEG memory diagnosis will be arrived through the blinded review of the EEG data

SECONDARY OUTCOMES:
The Montreal Cognitive Assessment (MoCA) performance | baseline
  This neuropsychological test will be used for cognitive screening. The scores on this test ranges from 0 to 30, and lower scores indicate decreased cognitive ability.
Mini Mental State Examination (MMSE) | baseline
  This neuropsychological test will be used to assess cognitive functioning. MMSE scores range from 0 to 30 with lower scores indicating decreased cognitive ability.
Consortium to Establish a Registry in Alzheimer's disease Word List Test (CERAD) | baseline
  The CERAD evaluates the immediate recall of a list of words (up to 30 correct recall on 3 individual recall trials), delayed recall (up to 10 correct recall after a 5 minute delay), and on yes-no recognition memory (up to 10 correct recognition)
Verbal Fluency test: Phonemic Test and the Category Fluency test | baseline
  Phonemic word fluency and categoric word fluency will be assessed using the Verbal Fluency: Phonemic Test and the Category Fluency test. For letter fluency, individuals name as many words as possible in one minute that start with the letters F, A, and S. For category fluency, individuals name as many words as possible in one minute that are within the Animals, Vegetables, and Fruits categories.
Trails Making Test A and B | baseline
  The Trail Making Test Part A consists of connecting a series a numbers with a line in ascending order as quickly as possible (performance is timed, and the score is the time to complete the task). The Trail Making Test Part B consists of connecting a series of letters and numbers, alternating back and forth between them, as quickly as possible in ascending order (performance is timed, and the score is the time to complete).This test will be used to assess the central executive functioning.
Boston Naming Test | baseline
  This test consists of 15 line drawings, with a maximum score of 15 correct. It will be used to assess naming skills in speakers of multiple languages
EEG amplitude | baseline
  EEG amplitudes will be measured from the EEG data
EEG latency | baseline
  EEG latency will be measured from the EEG data

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Turk, MD, Principal Investigator — BU Chobanian & Avedisian School of Medicine; Andrew Budson, MD, Principal Investigator — BU Chobanian & Avedisian School of Medicine
Locations (1):
- BU Alzheimer Disease Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No